CLINICAL TRIAL: NCT06754345
Title: 68Ga-NK224 PET Imaging of PD-L1 Expression in Cancers
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMYY-2023KY146
Record Dates: First submitted 2024-12-24; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Tumor; PD-L1
Keywords: Tumor; PD-L1; PET/CT; diagnosis
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: 68Ga-NK224 PET/CT: Each participant receives a single intravenous injection of 68Ga-NK224, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-NK224 positron emission tomography/computed tomography (PET/CT) for the evaluation of PD-L1 expression in primary and/or metastatic tumors, compared with histopathological results.

DETAILED DESCRIPTION:
Participants with cancer underwent 68Ga-NK224 PET/CT for an initial assessment. Tumor uptake was quantified by the maximum standard uptake value (SUVmax) and mean SUV (SUVmean). In addition, the PD-L1 expression of lesions was confirmed by histopathological analyzing. The quantitative parameters of 68Ga-NK224 PET/CT were compared with histopathological result to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order);
* (ii) patients with newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report);
* (iii) patients who had scheduled 68Ga-NK224 PET/CT scans;
* (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions;
* (ii) patients with pregnancy;
* (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (i) adult patients (aged 18 years or order); (ii) patients with newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report); (iii) patients who had scheduled 68Ga-NK224 PET/CT scans; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The concordance between 68Ga-NK224 PET/CT and histopathological result in PD-L1 expression | 30 Days
  For 68Ga-NK224 PET/CT parameter, the maximum standard uptake value (SUVmax) is measured by defining a region of interest (ROI) around the primary tumor. For histopathological results, the level of PD-L1 expression is quantified as low (<1%), medium (1-49%), and high (>49%), respectively. Finally, Kruskal-Wallis test will be used to test the concordance between 68Ga-NK224 PET/CT and histopathological result in PD-L1 expression.

SECONDARY OUTCOMES:
Evaluate the intra- and inter- tumor heterogeneity | 30 Days
  To assess inter-tumor heterogeneity, a quantitative measure of intratumoral heterogeneity, the heterogeneity index (HI), was calculated by dividing SUVmax by SUVmean for each lesion. Differences in 68Ga-NK224 uptake related to inter-tumor heterogeneity (between primary tumors and metastatic lesions) were analyzed using the Mann-Whitney U test.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China